CLINICAL TRIAL: NCT06703502
Title: Investigating the Efficacy of an Online Binge Eating Disorder Group Intervention for Under 18s
Brief Title: Evaluation of Pilot Online Binge Eating Disorder Group (BEG) in Under 18s.
Status: Completed | Type: Observational
Sponsor: Coventry and Warwickshire Partnership NHS Trust (Other Government)
Collaborators: Birmingham Newman University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 320293
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Binge Eating Disorder
Keywords: group; adolescent
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The National Institute for Clinical Excellence recommends a cognitive behavioural therapy (CBT) group intervention for binge eating disorder in under-18s. However, there is limited current research in this population. The present study sought to evaluate a CBT group intervention for binge eating disorder in under-18s.

DETAILED DESCRIPTION:
Background and study aims: The National Institute for Clinical Excellence recommends a cognitive behavioural therapy (CBT) group intervention for binge eating disorder in under-18s. However, there is limited current research in this population. The present study sought to evaluate a CBT group intervention for binge eating disorder in under-18s.

Who can participate? Participants were recruited from the Coventry Warwickshire Partnership Trust's Children and Young People Eating Disorders Team (n=2).

What does the study involve: Participating in a group intervention and completing questionnaires (Eating Disorder Examination - Questionnaire (EDE-Q), Revised Children's Anxiety and Depression Scale (RCADS) Child and RCADS Parent) before the group, at the end of the group and a follow-up appointment, as well as a feedback form at the end of the group intervention.

What are the possible benefits and risks of participating:

* Benefits: Working towards recovering from binge eating disorder
* Risks: As with all therapy, there is a risk of distress due to the topics discussed. There is no more risk than any other group online therapy.

Where is the study run from: Online intervention for participants who are eligible and who are under the care of the RISE Eating Disorders Team within Coventry and Warwickshire NHS Partnership Trust.

When is the study starting and how long is it expected to run for: The study commenced on on 23rd May 2023. The group intervention ran from 20th June 2023 to 26th September 2023.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Binge Eating Disorder
* Under 18 prior to the group commencing
* Spoke English fluently

Exclusion Criteria:

* If they were underweight. This was measured by percentage median body mass index (%mBMI) as recommended by the Medical Emergencies in Eating Disorders guidelines (Royal College of Psychiatrists, 2022) for under 18s. As such, individuals were excluded if %mBMI was less than 95%
* If they had any physical illness serious enough to prevent the participant from engaging fully in the group and completing the in-between session work
* If they were pregnant
* If they had an eating disorder-induced physical health state requiring regular medical intervention by the nursing team
* If they presented a mental health state requiring stabilisation prior to participating in the group intervention according the assessment team
* If they regularly used alcohol and/or drugs
* If they repeatedly self-harmed to the point of requiring additional interventions
* If they had a living situation not conducive to the start of an intervention (ongoing or upcoming changes).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population for study were young people (under 18) that are receiving support from the RISE Eating Disorder Team in the Coventry and Warwickshire Partnership Trust with a diagnosis of binge eating disorder.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire | 23rd May 2023-26th September 2023
  The questionnaire is designed to assess the range, frequency and severity of behaviours associated with a diagnosis of an eating disorder.

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (RCADS) Child | 23rd May 2023-26th September 2023
  The Revised Children's Anxiety and Depression Scale (RCADS) measures the reported frequency of various symptoms of anxiety and low mood.
Revised Children's Anxiety and Depression Scale (RCADS) Parent/Carer | 23rd May 2023-26th September 2023
  The Revised Children's Anxiety and Depression Scale (RCADS) measures the reported frequency of various symptoms of anxiety and low mood.
Feedback form | 23rd August 2023
  Feedback form asking questions about experience of the group and any recommendations for future groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Wood End Health Centre, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small population size, it does not feel appropriate to share the data.

DOCUMENTS (4):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT06703502/Prot_000.pdf
  • Informed Consent Form: Service User (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06703502/ICF_001.pdf
  • Informed Consent Form: Parent Carer version (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06703502/ICF_002.pdf
  • Informed Consent Form: 16+ Service User (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT06703502/ICF_003.pdf